CLINICAL TRIAL: NCT06632626
Title: Task-oriented Training on Hand Function in Patients With Taxanes-induced Peripheral Neuropathy
Brief Title: Task-oriented Training on Hand Function in Taxanes-induced Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Arwa Reda Hashem, Physical Therapy Specialist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/00460
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Neuropathy; Chemotherapy Effect; Hand Function
Keywords: Breast cancer; hand dexterity; hand grip strength; task-oriented training; Taxanes-induced peripheral neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Single-blind, randomized, controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Task oriented training group (Experimental): This group included 30 patients suffering from taxanes induced peripheral neuropathy who received 30 minutes of task-oriented exercises, three sessions per week for four weeks along with 30 minutes of the traditional physical therapy.
  Interventions: Other: Task oriented training exercises; Other: Traditional physical therapy
- Traditional physical therapy group (Active Comparator): This group included 30 patients suffering from taxanes induced peripheral neuropathy who received 30 minutes of the traditional physical therapy only, three sessions per week for four weeks.
  Interventions: Other: Traditional physical therapy

INTERVENTIONS:
Other: Task oriented training exercises — Task oriented training is a type of exercises in form of tasks using papers, pens, scissors, clips, coins, screws and clay
  Arms: Task oriented training group
Other: Traditional physical therapy — Traditional physical therapy inform of mobilization, strengthening exercises of hand and streching exercises.

SUMMARY:
Chemotherapy based on taxanes is commonly used to treat breast cancer. However, chemotherapy-induced peripheral neuropathy (CIPN), a side effect of taxanes, impairs a patient's grip strength, hand dexterity, and upper extremity function which affects quality of life (QOL).

DETAILED DESCRIPTION:
Task-oriented training, a type of exercise where exercises are organized into tasks, concentrates on enhancing particular functional abilities through useful, goal-directed activities. So, the purpose of the study to explore the effectiveness of task-oriented training (TOT) on grip strength, hand dexterity and upper extremity function in patients with taxanes-induced peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients were females only.
* Their ages range from 35 to 65.
* All patients suffered from CIPN after using taxanes (anti-cancer agent causing neurotoxic effect).
* Diagnosis of CIPN was determined based on symptom history or the presence of stocking glove pattern "distal dysesthesias, pain and numbness" beginning after taxanes intake.
* All patients enrolled to the study had their informed consent.
* Patients suffer from affected brachial plexus.

Exclusion Criteria:

* Patients had pain or numbness in the upper extremity due to other reasons like trauma (fracture), CNS diseases (cerebral infarction), other diseases with neurological symptoms like (diabetes, rheumatoid arthritis or cervical myelopathy).
* Patients had bone, brain or spinal cord metastases.
* Patients who had history of psychiatric disorders like: depression and schizophrenia or cognitive decline that may hinder them from active participation in the study.
* Patients exhibited only acute neuropathy like in patients using oxaliplatin.

Exclusion Criteria:

* Patients had pain or numbness in the upper extremity due to other reasons like trauma (fracture), CNS diseases (cerebral infarction), other diseases with neurological symptoms like (diabetes, rheumatoid arthritis or cervical myelopathy).
* Patients had bone, brain or spinal cord metastases.
* Patients who had history of psychiatric disorders like: depression and schizophrenia or cognitive decline that may hinder them from active participation in the study.
* Patients exhibited only acute neuropathy like in patients using oxaliplatin

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biologically female patients only
Enrollment: 60 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Hand grip strength | At baseline and after four weeks of intervention.
  Hand grip strength (HGS) was measured in the dominant hand for each patient using The CAMRY dynamometer
Hand dexterity | At baseline and after four weeks of intervention.
  The nine-hole peg test was used to assess the hand dexterity
Hand function | At baseline and after four weeks of intervention.
  Each patient was asked to answer the questions of the six scales in the Arabic version of Michigan hand questionnaire (1- Overall hand function, 2-Activities of Daily Living, 3- Work performance, 4- Pain, 5- Aesthetics, and 6- Satisfaction with hand function)

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa M A Elsayeh, PhD, Principal Investigator — Cairo University
Locations (1):
- faculty of physical therapy, Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersen Hammond E, Pitz M, Shay B. Neuropathic Pain in Taxane-Induced Peripheral Neuropathy: Evidence for Exercise in Treatment. Neurorehabil Neural Repair. 2019 Oct;33(10):792-799. doi: 10.1177/1545968319860486. Epub 2019 Jul 25. PMID 31342880
- [Background] Andersen Hammond E, Pitz M, Steinfeld K, Lambert P, Shay B. An Exploratory Randomized Trial of Physical Therapy for the Treatment of Chemotherapy-Induced Peripheral Neuropathy. Neurorehabil Neural Repair. 2020 Mar;34(3):235-246. doi: 10.1177/1545968319899918. Epub 2020 Jan 24. PMID 31976819